CLINICAL TRIAL: NCT04418674
Title: Comparison of Analgesic Effectiveness of Intravenous Ketamine and Fentanyl for Spinal Anesthesia is Sitting Position in Patients With Proximal Femur Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jenny Bajracharya (Other)
Responsible Party: Sponsor-Investigator, Jenny Bajracharya, Department of Anesthesia, Principal Investigator, Junior resident, B.P. Koirala Institute of Health Sciences
Organization: B.P. Koirala Institute of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRC/1597/019
Record Dates: First submitted 2020-05-31; First posted 2020-06-05 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2020-06

CONDITIONS: Fracture of Proximal End of Femur
Keywords: Spinal anesthesia; Ketamine; Fentanyl
MeSH Terms: interventions — Ketamine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Ketamine Group: Ketamine 0.3mg/kg intavenously before changing the position from supine to sitting for subarachnoid block.
  Fentanyl group: Fentanyl 1.5mcg/kg intravenously before changing the position from supine to sitting position for subarachnoid block.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 0.4ml from one 1 ml ampule of 50mg ketamine will be diluted with 9.6ml NS to make a concentration of 2mg Ketamine in each ml in a 10 ml syringe.
  One 2ml ampule of 100mcg Fentanyl will be diluted with 8 ml NS to make a concentration of 10mcg in each ml in a 10ml syringe
  Ketamine and Fentanyl will be administered as clear fluid from a 10ml syringe labelled as Study drug, therefore, both the patient and investigator will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Patient will be given Ketamine 0.3mg/kg intravenously before sitting positioning for subarachnoid block.
  Interventions: Drug: Ketamine
- Fentanyl (Active Comparator): Patient will be given Fentanyl 1.5mcg/kg intravenously before sitting position for subarachnoid block.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Ketamine — in this group, patient will receive ketamine at 0.3mg/kg intravenously.
  Arms: Ketamine
Drug: Fentanyl — In this group, the patients will receive fentanyl at 1.5mcg/kg intavenously.
  Arms: Fentanyl

SUMMARY:
This is a prospective comparative study which will be conducted in patients with proximal femur fracture undergoing operative interventions under subarachnoid block in sitting position. Ketamine group will receive 0.3mg/kg intravenously and Fentanyl group will receive 1.5mcg/kg before changing the position from supine to sitting for subarachnoid block. Analgesic effectiveness of the two drugs will be compared by Numeric Rating Scale for pain.

Research hypothesis (Null hypothesis) There is no difference in analgesic effectiveness, patient satisfaction, spinal performance and occurrence of adverse effects between Intravenous ketamine and intravenous fentanyl in patients with proximal femur fracture.

Alternate hypothesis Intravenous Ketamine in patients with proximal femur fracture improves the level of analgesia, patient satisfaction, spinal performance and occurrence of adverse effects when compared to intravenous fentanyl.

DETAILED DESCRIPTION:
Femur fracture is a common orthopedic problem following trauma in patients of all ages. It is a painful bone injury and is associated with severe pain and distress during preoperative period. Surgical repair is most commonly done in subarachnoid block. However, moving the patient for optimal positioning for spinal needle placement in subarachnoid space leads to severe pain. Adequate analgesia not only improves patient's comfort but has also been shown to improve positioning for subarachnoid block. Several analgesic modalities have been used to decrease movement evoked pain in these patients including the use of intravenous analgesics and blocks. However, there are only few studies comparing intravenous analgesics that alleviated the pain that occurs when changing position for subarachnoid block.

Patient enrollment will be done by the primary investigator one day prior to the surgery. All eligible patients with American Society of Anesthesiologist Physical Status I, II fulfilling the inclusion criteria will be informed about the study and written consent will be obtained in pre operative visit, one day prior to the surgery, in the orthopedic in-patient ward.

All patients will be kept nil per oral for 6 hours for solid, heavy meal, 4 hours for light meal and 2 hours for clear liquid. All the patients will be pre-medicated with Tab Lorazepam 1mg (<50kg) and 2mg (>50kg) orally the night before and in the morning of the surgery.

On the day of surgery, randomization will be done in pre operative holding area and the patient will be transferred to the operation theatre in trolley maintaining the skeletal traction. All standard monitoring devices like electrocardiogram, non-invasive blood pressure monitoring and pulse oximeter will be attached. Standard anesthesia monitoring including 3-lead electrocardiography, oxygen saturation(Spo2), blood pressure(BP) and heart rate(HR) will be done.Baseline Numeric Rating Scale(NRS) for pain at rest and movement will be assessed (movement is defined at 5 cm active vertical movement of the limb).

An intravenous line will be secured with 18 gauge intavenous cannula in the dorsum of hand. Pre-hydration will be started with Ringer's Lactate solution at 5ml/kg/hour.

Dose of the drug required according to the body weight will be calculated and prepared by the anesthetist not involved in the study. It will be labelled as study drug and will be delivered by the investigator.

Group A will receive Inj Ketamine 0.30mg/kg bolus dose. Group B will receive Inj Fentanyl 1.5mcg/kg bolus dose. The drug will be prepared in an identical sterile syringe as a clear fluid and will be labelled as "study drug".

Patient will receive the study drug according to randomization.Then, 10 minutes after delivery of the study drug, the patients will be kept in sitting position with the help of operation theatre assistant while maintaining the skeletal traction. Numeric Rating Scale will be enquired and noted. If the patient will report Numeric Rating Scale of 5 or more during placement in the sitting position, procedure will be stopped and fentanyl 20 microgram will given intravenously in the form of rescue analgesia before attempting to reposition again. Once the patient will be in sitting position subarachnoid will be performed in L 3-4 inter space using 2.4ml of 0.5% hyperbaric bupivacaine maintaining strict asepsis. The patient will be laid down back to supine position. The level of sensory block and motor block will assessed. After ascertaining adequate block, patient will be shifted to fracture table for operation. The number attempts required for successful subarachnoid block will be noted. The quality of patient positioning will subjectively be rated as good, satisfactory and optimal depending upon the ease of positioning for subarachnoid block by the anesthetist. Sedation scoring will be noted for 30 minutes after delivery of the study drug. All the vital parameters will be monitored continuously and recorded every 3 minutes for first 15 minutes then every 10 minutes throughout the surgery and once in Post Anesthesia Care Unit. Patient will be assessed for the presence any adverse effect of the study drug throughout the surgery. The level of satisfaction regarding the analgesia during positioning will be questioned to the patient using Likert Scale in PACU. The time required for the patients to be discharged from PACU will be noted.

Data management Data handling- Data will be entered in Microsoft Excel 2016 and converted into Statistical package for social sciences (SPSS 11.5) for statistical analysis Coding-Alpha numerical code will be used Monitoring-Data will be entered after every day of work. Data will be reported to guide and co-guides every week.

Statistical Methods Collected data will be entered in Microsoft Excel 2010 and be converted into SPSS software 11.5 version for statistical analysis.

For descriptive statistics percentage, mean, Standard deviation, median, interquartile range will be calculated along with graphical and tabular presentation. For inferential statistics Chi square test, independent t test, Mann Whitney U test will be applied to find out the significant difference between Fentanyl and Ketamine with selected clinical and demographic parameter at 95% confidence interval where level of significance is considered p <0.05.

ELIGIBILITY:
1. Inclusion criteria:

   Patients undergoing Subarachnoid block for proximal fracture femur
   1. Age: above 18 years
   2. ASA PS I, II
2. Exclusion criteria:

   1. Refusal to participate in the study
   2. Other painful co- morbidities
   3. Allergy or any contraindication to study medication
   4. Any contraindication to subarachnoid block
   5. Analgesics 8 hours prior to performing sunarachnoid block
   6. Pathologic fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale for Pain | 1 to 20 minutes
  Level of analgesia for subarachnoid block in sitting position measured by Numeric Rating Rating Scale for pain. Scale ranges from 0 to 10, where 0 is no pain and 10 being maximum/ worst imaginable pain.

SECONDARY OUTCOMES:
Likert Satisfaction score | 1 to 20 minutes
  Patient satisfaction for positioning the patient for subarachnoid block using Likert score will be used. It ranges from 1 to 5 (1=strongly dissatisfied, 2=dissatisfied, 3=neutral, 4=satisfied, 5=strongly satisfied)
Anesthetist Satisfaction Score | 1 to 20 minutes
  Anesthetist satisfaction for positioning the patient for subarachnoid block as good, satisfactory and Optimal
Number of attempts for successful spinal needle placement | 1 to 20 minutes (While performing subarachnoid block)
  Number of attempts for successful spinal needle placement
Adverse effects | 1 to 120 minutes (Intraoperatively)
  Occurrence of any adverse events like hypotension, bradycardia, hallucination, nausea and vomiting.
Modified Wilson Sedation Scale | 1 to 120 minutes (Intraoperatively)
  Sedation score of the patients will be noted (1=Oriented, 2=Drowsy,3=Arousable,4=Unarousable)
Modified Aldrerte Score | 10 to 30 minutes (In post anesthesia care unit)
  Time required by patients of each group to be discharged from the PACU will be noted bu using Modified Aldrerte Score (Score of 9-10=can be discharged, 8 or less=close monitoring needed)

CONTACTS AND LOCATIONS:
Overall Officials: Bishnu Pokharel, MS, Study Chair — B P Koirala Institute of Health and Sciences
Locations (2):
- Nepal (2):
  - B P Koirala Institute of Health and Sciences, Dharān, Sunsari
  - B P Koirala Institute of Health and sciences, Dharān, Sunsari

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diakomi M, Papaioannou M, Mela A, Kouskouni E, Makris A. Preoperative fascia iliaca compartment block for positioning patients with hip fractures for central nervous blockade: a randomized trial. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):394-8. doi: 10.1097/AAP.0000000000000133. PMID 25068412
- [Background] Sia S, Pelusio F, Barbagli R, Rivituso C. Analgesia before performing a spinal block in the sitting position in patients with femoral shaft fracture: a comparison between femoral nerve block and intravenous fentanyl. Anesth Analg. 2004 Oct;99(4):1221-1224. doi: 10.1213/01.ANE.0000134812.00471.44. PMID 15385380
- [Background] The safety, benefits and effectiveness of different intravenous subanesthetic doses of ketamine when combined with small dose of midazolam before combined spinal epidural technique for Orthopedic Lower Extremity Surgery Moataz Moataz Morad El-Tawil Anesthesia Department, Faculty of Medicine, Menoufya University Abstract
- [Background] Aral A Mohammed, MD*, Mayada M Ali, MD.Ketamine analgesia before spinal anesthesia for fractured femur. Sudan Med J 2015;April;51(1)